CLINICAL TRIAL: NCT06307990
Title: Advancing Understanding, Diagnosis and Monitoring of Thyroid Hormone Action Defects (ADAM-THAD)
Brief Title: Understanding, Diagnosis and Monitoring of Thyroid Hormone Action Defects
Acronym: ADAM-THAD
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: ASST Fatebenefratelli Sacco (Other); Federico II University (Other)
Responsible Party: Sponsor
Other Study IDs: 05M202
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Resistance, Thyroid Hormone
MeSH Terms: conditions — Thyroid Hormone Resistance Syndrome | interventions — Serologic Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — dried blood spots (DBS) peripheral blood cells extracted DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RTH Syndromes: Patients with THRA or THRB gene mutations
  Interventions: Genetic: NGS sequencing; Diagnostic Test: serological tests

INTERVENTIONS:
Genetic: NGS sequencing — analysis of candidate genes for RTHs syndromes, transporters defects or gene involved in thyroid hormone metabolism. Whole exome sequencing (WES) in a minority of cases
Diagnostic Test: serological tests — assessment of T4, T3 and other TH metabolites (LC-MS) in serum and dried blood spots

SUMMARY:
The goal of this observational study is to learn about the neurological and cardiological phenotype of patients with resistance to thyroid hormone (RTH) syndromes beta and alpha (RTHß and RTHa) due to dominant negative variants in the genes encoding the thyroid hormone receptors alpha (THRA) and beta (THRB).

The main question[s] it aims to answer are:

* Define frequency and improve early diagnosis for RTH syndromes
* Developing tools to accelerate diagnosis of RTH syndromes
* Development and validation of monitoring tools

Participants, recruited at neonatal screening or from cohorts of patients with unexplained specific neuro-cognitive or cardiovascular phenotypes will be submitted to biochemical and genetic investigations. In addition pluripotent stem cells will be generated from peripheral blood cells of RTHs patients and studied in vitro to understand the molecular mechanisms underlying neurological and cardiovascular consequences. In vitro and clinical data, will be correlated to identify biomarkers for monitoring treatment.

DETAILED DESCRIPTION:
TH action defects (THAD) are a group of rare syndromes characterized by abnormal thyroid hormone (TH) cell signaling due to defective transport, metabolism or action of TH via binding with nuclear receptors (TRs): there are two TRs, the alpha (TRa) and beta (TRß) receptors. Among them, mutations of THRA or THRB genes cause two distinct syndromes with Resistance to Thyroid Hormone (RTH) action whose incidence was estimated 1:20,000-50,000 newborns, likely representing the most frequent THAD forms. RTHa is due to dominant negative (DN) heterozygous mutations in THRA and characterized by dramatic manifestations in TRa-expressing tissues resembling untreated congenital hypothyroidism (CH).

RTHß is due to DN heterozygous THRB mutations, which cause variable TH resistance in TRß-expressing tissues (hypothalamus, pituitary, liver), resulting in distinctive biochemical signature (high free TH and unsuppressed TSH) together with additional features like deafness, impaired color vision and thyrotoxic-related symptoms (goiter, tachyarrhythmias, osteoporosis, anxiety and Attention-Deficit/Hyperactivity Disorder, ADHD).

Outstandingly, early treatment with TH or its analogues is expected to reduce most of the adverse consequences of RTHs but early/neonatal diagnosis is presently not feasible due to the lack of accurate biomarkers. Indeed, uniform characterization is essential for a rare disease, and establishment of clear-cut endocrine fingerprints for RTHa and RTHß are essential for a timely diagnosis.

In addition, the wide application of next generation sequencing (NGS) has yielded an unprecedented wealth of genetic information, calling for proper instruments to distinguish benign from pathogenic variants.

Finally, biomarkers for monitoring treatment of these conditions have not been established or validated.

This study aim to:

1. develop neonatal screening strategies for THAD and give unprecedented epidemiological characterization of RTHs in Italy
2. understand the pathogenicity of newly discovered THRB or THRA variants in in vivo model or identify new mechanisms
3. generate induced pluripotent stem cells from RTH patients to understand the molecular mechanisms underlying neurological and cardiovascular consequences and correlate in vitro and clinical data, with the final goal to identify potential biomarkers for monitoring treatment of these rare diseases.

ELIGIBILITY:
Inclusion Criteria:

- biochemical signature suggestive of RTHs syndromes at birth (a) or symptoms suggestive of RTHs syndromes (b) or known diagnosis of RTHs syndromes (c)

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Newborn patients (a) with normal TSH, but T3 and other TH metabolites suggestive of RTH syndromes, we will be submitted to genetic analysis
  Cohorts of patients (b) with unexplained: i) mental retardation and delayed development or epilepsy (ii) autism spectrum disorders (iii) growth maturation defects (iv) early onset cardiovascular diseases (v) with inappropriate tachycardia (vi) with ADHD or learning disorders (vii) early onset tachyarrhythmias, will be submitted to genetic analysis
  Patients with RTH syndromes already diagnosed and followed in the collaborating centers
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of Newborns With Abnormal Thyroid Hormone Levels Suggestive of Resistance to Thyroid Hormone (RTH) Syndromes, as Measured in Dried Blood Spots (DBS). | two years
  Thyroid hormone levels determinations in DBS of newborns
Frequency of Phenotypic Changes in Zebrafish Zygotes Microinjected with Human TR Variants, as a Measure of the Functional Impact of THRA and THRB Variants of Uncertain Significance (VUS). | two years
  Functional impact of THRA and THRB variant of uncertain significance (VUS) in the zebrafish model microinjected with different human TR variants
Direct differentiation of THRA mutant patients-derived human induced pluripotent stem cells (hiPSCs) to neural progenitors (hiPSc-CNeu) and cardiomyocyte (hiPSC-CMs) | two years
  Molecular characterization and electrophysiological characterization of hiPSc-CNeu and hiPSC-CMs carrying THRA and THRB variants and comparison with matched controls
To identify TH-target genes involved in determining stemness, proliferation potential and differentiation of hiPSC | two years
  Transcriptome analysis of hiPSc-CNeu and hiPSC-CMs

SECONDARY OUTCOMES:
Prevalence of Resistance to Thyroid Hormone (RTH) Syndromes in Specific Cohorts of Patients with Unexplained Phenotypes | two years
  To search novel RTHa cases in cohorts of patients with unexplained: i) mental retardation and delayed development or epilepsy (ii) autism spectrum disorders (iii) growth maturation defects (iv) early onset cardiovascular diseases. For RTHß, we aim to screen patients (i) with inappropriate tachycardia (ii) with ADHD or learning disorders (iii) early onset tachyarrhythmias.
Generation of a comprehensive RTH database | two years
  To establish a comprehensive RTH database including whole clinical/genetic/biochemical data of RTH patients, in view of the generation of a disease registry.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Istituto Auxologico Italiano IRCCS, Milan
  - Department of Endocrine & Metabolic Diseases, San Luca Hospital, Milan